CLINICAL TRIAL: NCT01581047
Title: Pharmacokinetics of Small Spectrum Beta-lactam Antibiotics (Amoxicillin/Clavulanic Acid and Cefuroxime) in Patients on Intensive Care Units
Acronym: AMOCEF
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/078; 2011-006107-35 (EudraCT Number)
Record Dates: First submitted 2012-02-15; First posted 2012-04-19 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Infection
Keywords: amoxicillin; clavulanic acid; cefuroxime; Patients in the intensive care unit, with an infection which requires amoxicillin/clavulanic acid or cefuroxime
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 8 serum samples will be taken per patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amoxicillin/Clavulanic Acid: Patients in the intensive care unit, with an infection which will be treated with Amoxicillin/Clavulanic Acid.
- Cefuroxime: Patients in the intensive care unit, with an infection which will be treated with Cefuroxime.

SUMMARY:
Adequate antibiotic therapy is very important in the treatment of infections. Spectrum and dosing of the antibiotics are two factors of the therapy: the spectrum of an antibiotic can't be changed, but the dosing scheme can be optimized. Recent studies proved that an optimized dosing scheme can improve the efficacy of the treatment. Broad-spectrum antibiotics have unpredictable pharmacokinetics in patients on intensive care units. This is due to the pathophysiologic processes in the patients on intensive care units: increased distribution volume, hypoproteinemia, organ failure… The investigators guess that similar processes influence the pharmacokinetics of small spectrum antibiotics (like amoxicillin and cefuroxime), but data lacks. Because the pharmacokinetics of broad spectrum antibiotics in seriously ill patients are better known, physicians are more confident prescribing these drugs. Studying the pharmacokinetic interactions of small spectrum antibiotics in seriously ill patients, can help to give the physician the confidence to prescribe these small-spectrum antibiotics.

In this study, the investigators will study the pharmacokinetics of amoxicillin/clavulanic acid and cefuroxime, in 60 patients on intensive care. 8 blood samples will be drawn via a central catheter on different moments after one administration of the antibiotic in the steady state phase. All the patients are prescribed the antibiotics for the treatment of their infections: they get the antibiotic therapy anyway. By measuring the concentrations on different moments after one administration, the investigators can reconstruct the pharmacokinetic function.

ELIGIBILITY:
Inclusion Criteria:

* patients on the intensive care unit, who are treated with amoxicillin/clavulanic acid or cefuroxime for an infection

Exclusion Criteria:

* informed consent lacking
* haematocrit < 21 %
* arterial catheter lacking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the intensive care unit, with an infection (which requires amoxicillin/clavulanic acid or cefuroxime).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2014-01-21 (Actual); Study Completion 2014-05-07 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) of Amoxicillin/Clavulanic acid. | Before and at 15, 30, 45, 60, 120, 240 and 360 minutes after administration
  The concentrations of the antibiotic in serum samples, drawn at various times after one administration, will be measured. With these data, we can calculate the time above the minimal inhibitory concentration (MIC).
Area under the serum concentration versus time curve (AUC) of Cefuroxime. | Before and at 15, 30, 45, 60, 120, 240 and 480 minutes after administration
  The concentrations of the antibiotic in serum samples, drawn at various times after one administration, will be measured. With these data, we can calculate the time above the minimal inhibitory concentration (MIC).

SECONDARY OUTCOMES:
Severity of disease classification. | At date of admission (day 1) and dismissal (up to 3 months).
  This will be assessed using the Acute Physiology and Chronic Health Evaluation II (APACHE2)-score.
Rate of organ failure. | At date of admission (day 1) and dismissal (up to 3 months).
  This will be assessed using the Sequential Organ Failure Assessment score (SOFA-score).
Concentration serum creatinin | At day 1.
24 hour urine creatinine clearance | At 24 hours
  Urine will be collected during 24 hours to measure the urine creatinine clearance.
Change in fluid balance | From 0 to 24 hours.
  Change in fluid balance will be measured.
Concentration serum albumin | At day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Waele, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium